CLINICAL TRIAL: NCT00167323
Title: Early Recovery Adherence Therapy for Bipolar Alcoholics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0307095
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2008-05-19 (Estimated); Status verified 2008-05

CONDITIONS: Bipolar Disorder; Alcohol Use Disorder
Keywords: Bipolar; Alcoholism
MeSH Terms: conditions — Bipolar Disorder; Alcoholism

INTERVENTIONS:
Behavioral: Adherence therapy

SUMMARY:
Effective psychosocial interventions for individuals with an alcohol use disorder co-occurring with a severe mental health problem such as bipolar disorder are lacking. Treatment engagement, adherence, and retention are a major challenge and crucial to achieving a favorable outcome. The early phase of recovery is a key period during which an effective intervention exerts its most significant impact. Our proposed treatment intervention is aimed at addressing early recovery issues, engagement, and treatment and medication adherence in bipolar alcoholics.

We propose to develop and refine a theoretically based and procedurally specified individual adherence therapy intervention for co-occurring alcohol use and bipolar disorder in early recovery, to develop standardized procedures, methods, and techniques so that treatment is delivered with a high degree of fidelity and competence, and to test the efficacy of this intervention through a randomized, parallel-group design comparing this new intervention with current regular clinical care.

DETAILED DESCRIPTION:
Co-occurring alcoholism and bipolar disorder is a significant comorbid condition representing serious clinical challenges and treatment difficulties and is associated with severe disabilities, morbidity, and heightened risk for suicide. Despite the recent increased attention to the problem of psychiatric comorbidity with alcoholism and other substance use disorders, little research has been conducted on this complex form of comorbidity, especially in regard to effective treatment approaches.

Enhancing treatment engagement, adherence, and retention is perhaps the most challenging clinical concern faced by clinicians caring for this population. Poor adherence is a major clinical problem among bipolar disorder with alcoholism. Poor adherence is associated with substantial medical expenses and loss of productivity.

Factors interfering with treatment adherence range from access to treatment, to health care providers disposition towards these patients, and to symptoms related to both bipolar disorder and alcoholism. Enhancing motivation for treatment and improving treatment adherence are essential components for an initial treatment intervention for this population. Our proposed treatment intervention is based on the principles of Motivational Enhancement Therapy and also integrates psychosocial and pharmacotherapy interventions that have been successfully used with alcoholism and other addictive disorders. It is practical and easy to learn and administer in the framework of general clinical care by health professionals with varied educational backgrounds.

ELIGIBILITY:
Inclusion Criteria:

1. Meet DSM-IV diagnostic criteria for Bipolar disorder and alcohol use disorder
2. Actively abusing alcohol (drinking on 2 or more occasions per week or having 3 or more drinks per occasion)
3. Have been stabilized on a mood stabilizer such as Valproate
4. Absence of any exclusion criteria

Exclusion Criteria:

1. Schizophrenia,, schizoaffective disorder or any psychotic disorder, unipolar major depression,, mental retardation, and signs of impaired cognitive functioning.
2. Any severe or unstable neurological and medical condition including epilepsy, history of brain injury, encephalitis, or any organic brain syndrome, severe cardiac, liver, kidney, endocrine, hematological, or impending surgery.

   Inability to read or understand the study forms and consent form
3. Pregnancy

The presence of non-alcohol substance use disorders will not constitute exclusion criteria unless it is clearly the drug of choice or it requires medications such as opioid substitution

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2003-07; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The proposed intervention with have:
A higher rate of treatment completion,
A higher rate of treatment adherence as indicated by the number of sessions attended,
An improved outcome as indicated by a higher percentage of alcohol free days, less average number of drinks per drinking days, longer period to relapse to heavy alcohol use, and greater improvement in their manic or depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ihsan M Salloum, MD, MPH, Principal Investigator — University of Pittsbugh
Locations (1):
- UPMC Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States